CLINICAL TRIAL: NCT05590871
Title: 3D Cardiac Electrophysiological Mapping System on Renal Artery Radiofrequency Ablation System for Hypertension: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: FlashPoint Renal Denervation Under Columbus 3D Mapping System Guidance for Treating Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Hongdian Medical CO., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 714156A
Record Dates: First submitted 2022-10-19; First posted 2022-10-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Renal Denervation (Experimental): Percutaneous renal denervation using the FlashPoint radio-frequency ablation system under the Columbus 3D mapping system guidance
  Interventions: Device: FlashPoint renal denervation system
- sham (Sham Comparator): For those subjects randomized to the sham procedure, renal artery angiography will serve as the sham procedure.
  Subjects maintenance of anti-hypertensive medications.
  Interventions: Other: Sham

INTERVENTIONS:
Device: FlashPoint renal denervation system — Radio-frequency ablation of renal arterial sympathetic nerves
  Arms: Renal Denervation
Other: Sham — After a renal angiography according to standard procedures, subjects remain blinded and remain on the catheterization lab table for at least 20 minutes prior to introducer sheath removal.
  Arms: sham

SUMMARY:
To verify the safety and effectiveness of the renal artery radiofrequency ablation system under the guidance of the three-dimensional cardiac electrophysiological mapping system in the renal denervation of essential hypertension.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, randomized controlled clinical study to verify the safety and efficacy of the renal artery radiofrequency ablation system under the guidance of the three-dimensional cardiac electrophysiological mapping system in the application of renal denervation of essential hypertension，designed to include drug-control research and sham-control resarch. Provide the basis for product registration and marketing and clinical application. Drug-control research include 65 subiects (5 are subjects trained and taught by the experimental group leader unit center, 40 subjects are randomly to the renal artery ablation with durg treatment group, 20 subjects to the drug treatment group). Sham-control research include 180 subjects, will be randomly assigned according to 2:1 (120 subjects in the renal artery ablation with drug treatment group and 60 subjects in the sham procedure with drug treatment group).

Patients will be followed for blood pressure measurement and antihypertensive medication at 1 month, 2 months, 3 months, 4 months, 5 months, 6 months, and 12 months after the procedure. Patients' urine samples will be collected for drug testing (LC-MS/MS) to determine their medication compliance in an independent laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 and ≤70 (not pregnant, breastfeeding, and have no reproductive plan within one year);
* Patients with essential hypertension, antihypertensive drug intolerance, and willing to undergo surgical treatment;
* Ambulatory blood pressure measurement 24-hour average systolic blood pressure ≥130mmHg or daytime ≥135mmHg, and pulse pressure difference <80 mmHg;
* A history of using antihypertensive medication within six months and blood pressure is still uncontrollable; standardized medication (at least two drugs) for at least 28 days before enrollment, and medication compliance ≥ 80%, office systolic blood pressure (OSBP) ) ≥ 150 mmHg and <180 mmHg, diastolic blood pressure (DBP) ≥ 90 mmHg;
* The patients agree to participate in this clinical trial and sign the informed consent form, agreeing to follow-up evaluation under the requirements of the verification protocol.

Exclusion Criteria:

* Renal artery anatomy failures include:

  1. Renal artery diameter <4mm or treatment length <20mm;
  2. Renal artery stenosis >50% or renal aneurysm on either side;
  3. A history of renal artery intervention, including balloon angioplasty or stenting or RDN;
* Glomerular filtration rate (eGFR) <45mL/min/1.73m2 (MDRD formula);
* History of hospitalization for hypertensive crisis in the past year;
* During the screening and lead-in period, the patient used antihypertensive drugs other than the standard antihypertensive drugs prescribed in this study protocol;
* Nocturnal sleep apnea syndrome requires mechanical ventilation (such as tracheostomy);
* Those who have or are currently suffering from the following diseases or conditions:

  1. Primary pulmonary hypertension (moderate to severe);
  2. Type I diabetes;
  3. History of any cerebrovascular events (eg, stroke, transient cerebral ischemic event, cerebrovascular accident) within 3 months;
  4. History of any serious cardiovascular event within 3 months (eg, myocardial infarction, CABG, acute heart failure requiring hospitalization (NYHA III-IV), unstable angina attack);
  5. Factors that interfere with blood pressure measurement in any case (eg, patients with severe peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, severe anemia);
  6. Arranged or planned surgery or cardiovascular intervention within the next 6 months;
  7. Patients with malignant tumors and end-stage diseases who survival period is less than 1year;
* Patients with secondary hypertension.
* Patients who are deemed inappropriate to participate in this trial by other investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
24-hour ambulatory mean systolic blood pressure reduction | Baseline to 6 months
  The primary effectiveness endpoint is change in 24-hour ambulatory mean systolic blood pressure from baseline to 6 months post-randomization
The incidence of Major Adverse Events (MAE) | Baseline to 1 month
  Safty outcome

SECONDARY OUTCOMES:
Reduction in office systolic and diastolic BP | Baseline to 1, 3, 6 months post procedure
  Secondary outcome
Reduction in average 24h ambulatory diastolic BP | Baseline to 1, 3, 6 months post procedure
Reduction in home systolic and diastolic BP | Baseline to 1, 2, 3, 4, 5, 6 months post procedure
Percentage of subjects change the number, class, dose of antihypertensive drugs | Baseline to 1, 2, 3, 4, 5, 6 months post procedure
Difference in antihypertensive drug burden index | Baseline to 6 months post procedure
Subjects level of TTR ( time in target BP range) | Baseline to 6 months post procedure
Success rate of the renal interventional therapy procedure | during the procedure
  Procedure success rate defined as successful introduction of the catheter, navigation to the treatment site, and there are no procedure-related SAE.
Incident of acute procedure safety events | 7 days post procedure
Incident of chronic procedure safety events | 6 months post procedure
Incidence of TTR with MAE, all cause death, stroke and myocardial infarction | Baseline to 6 months post procedure
Incidence of adverse events | Baseline to 6 months post procedure
Incident of serious adverse events | Baseline to 6 months post procedure
Ablation system defect rate | During procedure

CONTACTS AND LOCATIONS:
Locations (27):
- China (27):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - Cardiovascular Hospital Affiliated to Xiamen University, Xiamen, Fujian
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhenzhou, Henan
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Ansteel Group General Hospital, Anshan, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shengyang, Liaoning
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Weifang People's Hospital, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Air Force Medical University of PLA, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yan'an Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Shenzhen Guangming District People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No